## **IMPACT-AF SAP**

NOT FOR REPRODUCTION

NCT 01927367

# Optimizing primary care management of atrial fibrillation: The rationale and methods of the Integrated Management Program Advancing Community Treatment of Atrial Fibrillation (IMPACT-AF) study Statistical Analysis Plan, Version 1 January 9, 2019

#### **Background**

The burden of Atrial Fibrillation (AF), the most common sustained cardiac rhythm abnormality, is growing markedly such that the lifetime risk of acquiring this condition is now around 1 in 4.<sup>1,2</sup> AF is linked to increased mortality, substantial morbidity, high patient and health care costs,<sup>3</sup> as well as impaired quality of life.<sup>4</sup> In particular, AF is an important and independent risk factor for stroke, increasing the risk of such events by 5-fold and accounting for approximately 15-20% of all strokes.<sup>5</sup> Since at least a third of AF patients are asymptomatic,<sup>6</sup> many cases will be identified in outpatient settings when patients are being assessed for other conditions.

Traditionally, the major therapeutic interventions in AF patient care are directed at modifying or reversing the irregular rhythm and fast heart rate and in providing antithrombotic therapy to prevent strokes.<sup>7-9</sup>

Recently, multi-disciplinary approaches to AF management, centered on specialty AF clinics, have reported encouraging clinical results, including reductions in wait times for specialist assessment, emergency department (ED) visits, hospitalizations, and even mortality. However, such clinics require expert staff, broad collaboration, and special resources including physical space that entail high costs.

Clinical Decision Support Systems (CDSS) are intelligent systems that digitize and operationalize evidence-based guidelines, clinical pathways and algorithms to provide personalized, timely and evidence-informed functions. While the utility of such heath informatics approaches to health care might seem intuitive, this is not always the case. The diversity in the design, functionality and implementation of CDSS in real-life care settings has precluded making sweeping judgments about their clinical effectiveness, particularly over the longer term. While such technologies offer promise, more robust systems need to be developed and their effectiveness assessed, ideally in randomized trials.

We have developed a CDSS tool that aims to empower improvement in overall AF-related care, not simply with regards to antithrombotic management, but also to support effective rate control and treatment of AF risk factors. The tool has been assessed in a preliminary fashion by a general cardiologist, electrophysiologist and primary care physician, working independently to assess the

utility and dependability of the CDSS using mock clinical cases. While it functioned accurately and with seeming efficacy, there remains the need to determine applicability, ease of use and clinical effectiveness in terms of whether AF patient care and outcomes would improve at the population level with its use.

The primary aim of Integrated Management Program Advancing Community Treatment of Atrial Fibrillation (IMPACT-AF) study is to evaluate whether a CDSS tool, available to primary care physicians, and designed to support both practitioners and patients with evidence-based AF management, can improve clinical and patient-reported outcomes by comparison to usual clinical care. It further seeks to establish whether it will better standardize process of care so as to produce more efficient and cost-effective use of time and scarce health care resources as compared to usual care.

#### Methods

IMPACT-AF is a prospective, randomized, un-blinded, cluster design clinical trial, conducted in the primary care setting of Nova Scotia, Canada.

At least 200 primary care providers are being recruited and randomized at the level of the practice to control (usual care) or intervention (eligible to access to CDSS) cohorts. Over 1,000 patients of participating providers with confirmed AF will be managed per their provider's respective assignment.

#### Outcomes

#### Primary Outcome

The IMPACT-AF primary outcome is composite of any AF-related emergency department visit or unplanned CV hospitalization over 12 months.

#### Secondary Outcomes

Secondary outcomes include comparing the intervention versus usual care over 12 months on the following:

- 1. Any AF-related emergency department visit
- 2. Unplanned cardiovascular (CV) hospitalization
- 3. Strokes
- 4. Systemic embolism / major bleeding
- 5. Mortality
- 6. Anticoagulant therapy
- 7. Access to specialist consultation

- 8. Echo
- 9. Catheter ablations
- 10. EQ5D
- 11. Health care costs

The definitions of all outcome variables for the primary and secondary analyses are found in Appendix 1.

#### **Analysis Plan**

This statistical analysis plan follows the JAMA Guidelines for the Content of Statistical Analysis Plans in Clinical Trials <sup>13</sup>. A summary of all planned analyses is provided in **Table 1**.

#### Blinded Analyses

All statistical analyses will first be completed using blinded treatment groups (i.e. treatment X and Y).

#### Presentation of Data

The trial results will be presented according to the CONSORT guidelines for randomized controlled trials (RCTs)  $^{14}$ . The baseline demographic characteristics of the patients will be summarized by group, reported as a mean (standard deviation [SD]) or median (first quartile, third quartile) for continuous variables and count (percent) for categorical variables (**Tables 2**). All statistical tests will be 2-tailed with  $\alpha$ =0.05.

#### Primary Outcome Analysis

The primary efficacy analysis will be an analysis to compare rates of the composite of any AF-related emergency department visit or unplanned CV hospitalization between Intervention and Usual care over 12 months, with the outcome being treated as number of events (Tables 3). The analysis will follow the intention-to-treat (ITT) principle. While the unit of randomization is the practice/physician, the unit of analysis will be the patient. We will use Generalized Estimating Equations (GEE) —assuming exchangeable correlation structure for patients within the same practice and adjusting for urban and rural practice types to analyze all outcomes<sup>15</sup>. Unlike ordinary regression techniques, GEE allows us to estimate the intra-practice correlation among patients within each practice. For time-to-event analysis this is done using frailty-models. The results will be reported as estimate of the effect—reported as hazard ratio [HR], corresponding 95% confidence interval and associated p-values. All p-values will be reported to three decimal places with those less than 0.001 reported as p<0.001. The criterion for statistical significance will be set a priori at alpha = 0.05. The answers to the five questions in the EQ-5D-5L will be converted to health utilities using the Canadian scoring algorithm<sup>16</sup>. Cost effectiveness analysis

will be conducted by calculating the incremental cost per QALY gained by the CDSS arm compared with the usual care arm. Due to skewness of costs and health utility distributions, the non-parametric bootstrapping method will be used to estimate the 95% confidence interval for the incremental cost per QALY gained. All analyses will be performed using SAS version 9.4 (Cary, NC).

#### Secondary Outcomes Analysis

We will estimate the effect of CDSS (intervention) versus usual care (control) over 12 months on the following: any AF-related emergency department visit; unplanned CV hospitalization; strokes; systemic embolism / major bleeding; mortality; anticoagulant therapy; access to specialist consultation; echo; catheter ablations; EQ5D; health care costs (Table 3). The subgroup analyses will be performed by adding an interaction term of the subgroup variable and the intervention variable in the model. The criterion for statistical significance for subgroup analyses will be set at alpha = 0.05. This will not be adjusted for multiple testing as these analyses are exploratory.

#### Sensitivity Analyses

There are several methods for analyzing cluster RCTs<sup>17, 18</sup>. We will conduct sensitivity analyses in two ways. Firstly, we will perform sensitivity analyses using commonly used patient-level methods such as random-intercept model method (Table 4a). Secondly, we will also perform sensitivity analyses with the outcome (composite of any AF-related emergency department visit or unplanned CV hospitalization) being treated as a count assuming a Poisson distribution (Table 2). The results will be reported as incidence rate ratio [IRR], 95% CI and associated p-value. We hypothesize that our results will remain robust to the different sensitivity analyses.

#### Subgroup Analyses

A subgroup analysis will be conducted to compare the effect of CDSS (intervention) versus usual care (control) on the composite of any AF-related emergency department visit or unplanned CV hospitalization, as well as the of number AF Related ED Visits and CV Hospitalizations individually, by location of practice, patient sex, age, CHADS2, CHADS-VASC, hypertension, diabetes and years of practice of family doctor. We will perform these subgroup analyses by regression methods with appropriate interaction terms. This subgroup analysis will be conducted for all primary and secondary outcomes (Tables 5a, 5b and 5c). Our hypothesis is that the effects of the intervention on outcomes differ by subgroups. A sensitivity analysis will equally be conducted for all the different subgroup analyses with the outcome being treated as a count (Tables 5a, 5b and 5c). All the subgroup results will be presented using forest plots reporting estimates of effect as HR or IRR, 95% CI for each subgroup and a p-value of the interaction test.

#### Dissemination

Upon trial completion, the primary manuscript with the 12-month follow-up results, whether positive, negative or neutral, will be submitted for a peer-reviewed publication to a top medical journal. The final dataset will be shared through an open access data repository once all analyses are completed.

#### References

- 1. Ball J, Carrington MJ, McMurray JJ, et al. Atrial fibrillation: profile and burden of an evolving epidemic in the 21st century. Int J Cardiol 2013;167:1807-24.
- 2. Chugh SS, Havmoeller R, Narayanan K, et al. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation 2014;129(8):837-47.
- 3. Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jiménez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P. American heart association statistics committee and stroke statistics subcommittee. Heart disease and stroke statistics—2017 update: a report from the American Heart Association [published online ahead of print January 25, 2017]. Circulation. 2017;135(10):e146-603. https://doi.org/10.1161/CIR.00000000000000485. [Epub 2017 Jan 25].
- 4. Thrall G, Lane D, Carroll D, et al. Quality of life in patients with atrial fibrillation: a systematic review. Am J Med 2006;119(5):448.e1-448.e19.
- 5. Reiffel JA. Atrial fibrillation and stroke: epidemiology. Am J Med 2014;127:e15-6.
- 6. Savelieva I, Camm AJ. Clinical relevance of silent atrial fibrillation: prevalence, prognosis, quality of life, and management. J Interv Card Electrophysiol 2000;4(2):369-82
- 7. January CT, Wann LS, Alpert JS, et al. 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society Developed in Collaboration With the Society of Thoracic Surgeons. J Am Coll Cardiol 2014;64(21):e1-76.
- 8. Kirchhof P, Benussi S, Kotecha D, et al. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J 2016;37(38): 2893-962.
- 9. Verma A, Cairns JA, Mitchell LB, et al. 2014 focused update of the Canadian Cardiovascular Society guidelines for the management of atrial fibrillation. Can J Cardiol 2014;30:1114-30.

- 10. Gillis AM, Burland L, Arnburg B, et al. Treating the right patient at the right time: an innovative approach to the management of atrial fibrillation. Can J Cardiol 2008;24(3):195-8.
- 11. Hendriks JM, de Wit R, Crijns HJ, et al. Nurse-led care vs. usual care for patients with atrial fibrillation: results of a randomized trial of integrated chronic care vs. routine clinical care in ambulatory patients with atrial fibrillation. Eur Heart J 2012;33: 2692-9.
- 12. Hendriks JM, Crijns HJ, Vrijhoef HJ. Integrated chronic care management for patients with atrial fibrillation: a rationale for redesigning atrial fibrillation care. J Atr Fibrillation 2015;7(5):45-50.
- 13. Gamble C, Krishan A, Stocken D, Lewis S, Juszczak E, Dore C, Williamson PR, Altman DG, Montgomery A, Lim P, Berlin J, Senn S, Day S, Barbachano Y, Loder E. Guidelines for the content of statistical analysis plans in clinical trials. JAMA. 2017;318(23):2337-43.
- 14. 15. Schulz KF, Altman DG, Moher D, for the CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010;340:c332.
- 15. Hardin JW, Hilbe JM. Generalized estimating equations. New York, NY: Chapman & Hall/CRC. 2001.
- 16. Xie F, Pullenayegum E, Gaebel K, et al. A time trade-off value set of the EQ-5D-5L for Canada. Med Care 2016;54:98-105.
- 17. Ma J, Thabane L, Kaczorowski J, et al. Comparison of Bayesian and classical methods in the analysis of cluster randomized controlled trials with a binary outcome: the Community Hypertension Assessment Trial (CHAT). BMC Med Res Methodol 2009;9:37. https://doi.org/10.1186/1471-2288-9-37.
- 18. Diggle PJ, Liang K-Y, Zeger S. Analysis of Longitudinal Data. Oxford: Oxford Science Publications. 1994.
- 19. Briel M, Lane M, Montori VM, Bassler D, Glasziou P, Malaga G, Akl EA, Ferreira-Gonzalez I, Alonso-Coello P, Urrutia G, Kunz R, Culebro CR, da Silva SA, Flynn DN, Elamin MB, Strahm B, Murad MH, Djulbegovic B, Adhikari NKJ, Mills EJ, Gwadry-Sridhar F, Kirpalani H, Soares HP, Elnour NOA, You JJ, Karanicolas PJ, Bucher HC, Lampropulos JF, Nordmann AJ, Burns KEA, Mulla SM, Raatz H, Sood A, Kaur J, Bankhead CR, Mullan RJ, Nerenberg KA, Vandvik PO, Coto-Yglesias F, Schunemann H, Tuche F, Chrispim PPM, Cook DJ, Lutz K, Ribic CM, Vale N, Erwin PJ, Perera R, Zhou Q, Heels-Ansdell D, Ramsay T, Walter SD, Guyatt GH. Stopping randomized clinical trials early for benefit: a protocol of the study of trial policy of interim truncation-2 (STOPIT-2). Trials. 2009;10:49.

20. Montori VM, Devereaux PJ, Adhikari NK, Burns KE, Eggert CH, Briel M, Lacchetti C, Leung TW, Darling E, Bryant DM, Bucher HC, Schunemann HJ, Meade MO, Cook DJ, Erwin PJ, Sood A, Sood R, Lo B, Thompson CA, Zhou Q, Mills E, Guyatt GH. Randomized trials stopped early for benefit: a systematic review. JAMA. 2005;294:2203-9.

**Table 1: Statistical Analysis Plan Summary** 

| Objective | Outcome | Hypothesis | Methods of Analysis |
|---|---|---|---|
| 1) Primary To compare rates of the composite of any AF-related emergency department visit or unplanned CV hospitalization between Intervention and Usual care over 12 months | composite of any AF-related emergency department visit or unplanned CV hospitalization over 12 months | Intervention better than<br>Usual Care | Generalized Estimating<br>Equations (GEE) or frailty<br>models |
| 2) <u>Secondary</u> To compare I vs UC over 12 months on the following: any AF-related emergency department visit | any AF-related<br>emergency<br>department visit | Intervention better than<br>Usual Care | GEE or frailty models |
| unplanned CV<br>hospitalization | unplanned CV<br>hospitalization | Intervention better than Usual Care | GEE or frailty models |
| strokes | strokes | Intervention better than Usual Care | GEE or frailty models |
| systemic embolism / major<br>bleeding | systemic embolism /<br>major bleeding | Intervention better than Usual Care | GEE or frailty models |
| mortality | mortality | Intervention better than Usual Care | GEE or frailty models |
| anticoagulant therapy | anticoagulant<br>therapy | Intervention better than Usual Care | GEE or frailty models |
| access to specialist consultation | access to specialist consultation | Intervention better than Usual Care | GEE or frailty models |
| echo | echo | Intervention better than Usual Care | GEE or frailty models |

| catheter ablations | catheter ablations | Intervention better than | GEE or | frailty models |
|---|---|---|---|---|
| | | Usual Care | | |
| EQ5D | EQ5D | Intervention better than | GEE or | frailty models |
| | | Usual Care | | |
| health care costs | health care costs | Intervention better than | GEE or | frailty models |
| | | Usual Care | | |
| 3) Subgroup Analyses: | | | | |
| To compare the effect of I | | | | |
| vs UC by different | All primary and | Effects on outcomes | Regres | sion methods with |
| subgroups: location of | secondary outcomes | differ by location of | approp | riate interaction |
| practice, patient sex, | | practice | term | |
| age, CHADS2, CHADS- | | | | |
| VASC, hypertension, | | | | |
| diabetes and years of | | | | |
| practice of family doctor | | | | |
| 4) Sensitivity Analyses: | composite of any | Results will remain | i) | patient-level |
| i) To assess the robustness | AF-related | robust | | methods such as |
| of the results to different | emergency | | | random-intercept |
| methods of adjusting for | department visit or | | | model and |
| clustering; | unplanned CV | | | cluster-level [i.e. |
| ii) To assess the robust | hospitalization | | | random- and |
| ness of the results if the | | | | fixed-effects |
| outcome is treated as the | | | | meta-analytic] |
| count (number of events) | | | ii) | GEE using |
| | | | | Poisson |
| | | | | distribution |

#### **IMPORTANT REMARKS:**

- The GEE is a technique that allows to specify the correlation structure between patients within a hospital and this approach produces unbiased estimates under the assumption that missing observations will be missing at random. An amended approach of weighted GEE will be employed if missing observations are found not to be at random.
- In all analyses results will be expressed as coefficient, standard errors, corresponding 95% and associated p-values.
- Goodness-of-fit will be assessed by examining the residuals for model assumptions and chi-squared test of goodness-of-fit.

Table 2. Characteristics of the Study Populations at Baseline

| Characteristic | Variable | Usual<br>Care<br>(N=543) |
|---|---|---|
| Age – years<br>Median<br>Interquartile range | Age at start | |
| Male sex - n (%) | Sex (Male) | |
| Height – cm - Mean (SD) | Height | |
| Weight – Kg- Mean (SD) | Weight | |
| Urban location of care - n (%) | Location | |
| Heart rate – BPM - Mean (SD) | Heart Rate | |
| Systolic Blood pressure -<br>mmHg<br>Median<br>Interquartile range | Systolic BP | |
| Systolic Blood pressure -<br>mmHg<br>Median<br>Interquartile range | Diastolic BP | |
| Type of atrial fibrillation - n (%) | | |
| Paroxysmal | AF Classification (Paroxysmal) | |
| Persistent | AF Classification (Persistent/Chronic) | |
| Newly diagnosed/new onset | AF Classification (First Episode) | |
| PREVIOUS MEDICATION USE - n (%) | | |
| Aspirin | Ingredient (Aspirin) | |
| other antiplatelet | Ingredient (TICLOPIDINE) or (PRASUGREL) or (TICAGRELOR) or (CLOPIDOGREL) | |
| Vitamin K antagonist<br>(Warfarin) | Ingredient (Warfarin) | |
| Non-vitamin K antagonist (NOAC) | Ingredient (DABIGATRAN) or (RIVAROXABAN) or (APIXABAN) | |
| Beta-blocker | Ingredient (TIMOLOL) or (LABETALOL) or (CARVEDILOL) or (PINDOLOL) or (ACEBUTOLOL) or (PROPANOLOL) or (NADOLOL) or (ATENOLOL) or (BISOPROLOL) | |
| Calcium channel blocker | Ingredient (NIFEDIPINE) or (FELODIPINE) or (AMLODIPINE) or (AMLODIPINE + ATROVASTATIN) or (DILTIAZEM) or (VERAPAMIL) | |
| Digoxin | Ingredient (DIGOXIN) | |
| Any other antiarrhythmic | Ingredient (DRONEDARONE) or (QUINIDINE) or (PROCAINAMIDE) or (MEXILETINE) or | |

| | (SOTALOL) or (LIDOCAINE) or (FLECAINIDE) or (PROPAFENONE) or (AMIODARONE) |
|---|---|
| Nonsteroidal anti-<br>inflammatory | Ingredient (SULINDAC) or (PETOPROPHEN) or (PIROXICAM) or (KETOROLAC) or (TENOXICAM) or (TIAPROFENIC) or |
| | (INDOMETHACIN) and (ETODOLAC) or<br>(NEPAFENAC) or (IBUPROFEN) or |
| | (MELOXICAM) or (NAPROXEN) or<br>(DICLOFENAC) or (CELECOXIB) |
| OAC contraindication | OAC Contraindication (Yes) |
| OAC other reason not prescribed | OAC reason not Rxd (Yes) |
| BLEEDING AND STROKE RISK SCORES | |
| CHA <sub>2</sub> DS <sub>2</sub> | NOT the value REPORTED in PCP chart. |
| Score - Mean (SD)<br>Score - n (%) | CALCULATED using documented RFs. |
| 0 | |
| 1 2 | |
| 2 3 | |
| 4 | |
| 5 | |
| 6 | |
| 7<br>CHA <sub>2</sub> DS <sub>2</sub> -VASc | NOT the value REPORTED in PCP chart. |
| Score - Mean (SD)<br>Score - n (%) | CALCULATED using documented RFs. |
| 0 | |
| 1 | |
| 2 | |
| 3 4 | |
| 5 | |
| 6 | |
| 7 | |
| 8 9 | |
| Bleeding risk: HAS-BLED | |
| Score - Mean (SD) | |
| Score - n (%)<br>1 | |
| 2 | |
| 3 | |
| 4 | |
| 5 | |
| 6 | |

| 7 | |
|---|---|
| 7<br> 8 | |
| 9 | |
| COEXISTING CONDITIONS - n | |
| (%) | |
| Previous stroke, systemic | Stroke (Yes) or SE (Yes) or TIA (Yes) |
| embolism or transient | Stroke (163) of 3E (163) of 11A (163) |
| ischemic attack | |
| Congestive heart failure | HF/LV Dysfunction (Yes) |
| Hypertension | Hypertension (Yes) or (Yes-Treated) or (Yes- |
| rrypertension | Not Treated) |
| Diabetes mellitus | Diabetes (Yes-Not Documented) or (Yes-Type |
| Diabetes memeas | 1) or (Yes-Type 2) |
| Previous myocardial | MI (MM-YYYY) or (ND) |
| infarction | |
| Vascular disease (any) | Vascular Disease (Yes) |
| CAD | CAD (Yes) |
| PAD/PVD | Aortic Plaque (Yes) |
| UA | PAD/PVD (Yes) |
| MI | UA (date) (MM-YYYY) or (ND) |
| Aortic plaque | MI (date) (MM-YYYY) or (ND) |
| Valvular Heart Disease | Replacement Type (Mechanical) or Mitral |
| | Stenosis Type (Moderate) or (Severe) |
| Congenial Heart Disease | Congenital Heart Disease (Yes) |
| OSA | OSA Dx (Yes) |
| Tobacco use | |
| Former | Tobacco use (Former) |
| Current | Tobacco use (Current) |
| Alcohol abuse | Alcohol abuse (Yes) |
| Pericarditis | Pericarditis (Yes) |
| Pulmonary Disease | Pulmonary Disease (Yes) |
| INITEDVENITIONS (PROCEDURES | |
| INTERVENTIONS/PROCEDURES | |
| - n (%) | Vascular Procedure (Vas) |
| Vascular procedure (any) CABG | Vascular Procedure (Yes) CABG (Yes) |
| PCI | PCI (Yes) |
| Ablation (for flutter or AF) | AF Ablation (Yes) or Previous Ablation for Aflu |
| Ablacion (for naccer of All) | (Yes) |
| Pacemaker / ICD | Pacemaker (Yes) |
| Cardioversion | |
| # of patients | Cardioversion (Yes) |
| # of events – median (IQR) | Cardioversions no. |
| Bleeding History - n (%) | |

| Any bleeding | Bleeding History (Yes) |
|---|---|
| Intracranial | IC-Intracerebral (Yes) or IC-Other (Yes) |
| Non-intracranial | NIC-Epistaxis (Yes) or NIC-GI (Yes) or NIC- |
| Non intractation | Other (Yes) |
| Major bleeding | Major bleeding (Yes) |
| PAST REFERRALS - n (%) | major siecumg (res) |
| , , | |
| AF Clinic | Referred to (AF Clinic) |
| Cardiologist | Referred to (Cardiologist) |
| Internist | Referred to (Internist) |
| Electrophysiologist | Referred to (Electrophysiologist) |
| Cath ablation | Referred to (Cath Ablation) |
| ED visit for AF within the last | |
| 12 months | ER Visits (Yes) |
| # of patients - n (%) | ED Visits |
| # of events - Mean (SD) | 1 |
| | 2 |
| | 3 |
| | >3 |
| Cardiovascular-related | |
| hospitalization within the last | |
| 12 months | CV Hospitalization (Yes) |
| # of patients - n (%) | CV Hospitalizations |
| # of events - Mean (SD) | 1 |
| | 2 |
| | 3 |
| LAB VALUES | ) |
| eGFR – ml/min | Value when Blood Work (eGFR) |
| Median | |
| Interquartile range | |
| eGFR - n (%) | |
| < 30 ml/min | |
| 30-50 ml/min | |
| > 50 ml/min | |
| Hemoglobin - g/L | Value when Bloodwork (Hemoglobin) |
| Median | value when bloodwork (Hemoglobin) |
| Interquartile range | |
| Platelet - µmol/L | Value when Bloodwork (platelet count) |
| Median | value when bloodwork (platelet county |
| Interquartile range | |
| TSH - mIU/L | Value when Bloodwork (TSH) |
| Median | Talle William Blood Work (1911) |
| Interquartile range | |
| INR | |
| CARDIAC ASSESSMENTS | |
| Prior ECHO - n (%) | ECHO (Yes) |
| Ejection Fraction | The calculated EF |
| Licetion Fraction | THE CARCUIATED ET |

| Patients with EF - n (%) | |
|-----------------------------|----------------------------|
| EF -Mean (SD) | |
| Normal (≥ 51%) | |
| Slightly Reduced (41-50%) | |
| Moderately Reduced (31-40%) | |
| Severely Reduced (≤ 30%) | |
| Stress Test | Stress Test (Yes) |
| Holder or Loop - n (%) | Holter (Yes) or Loop (Yes) |
| ECG within 12 months | ECG (Yes) |

Table 3. Primary and Secondary outcomes at 12-months

| Outcome<br>(Usual Care is reference) | Interventio<br>(N= | - | Gro | (N=) analysis an | | Sensitivity<br>analysis |
|---|---|---|---|---|---|---|
| | No. of<br>Patients | No. of<br>Events | No. of Patients | No. of<br>Events | HR (95% CI);<br>p-value | IRR (95% CI),<br>p-value |
| Primary | | | | | | |
| AF related ED visits or CV hospitalizations | | | | | | |
| Secondary | | | | | | |
| AF related ED visits | | | | | | |
| Heart Failure | | | | | | |
| Syncope/Presyncope | | | | | | |
| TIA/Stroke | | | | | | |
| ACS (UA/MI) | | | | | | |
| Rate/Rhythm | | | | | | |
| Unplanned CV | | | | | | |
| hospitalization | | | | | | |
| Heart Failure | | | | | | |
| Syncope/Presyncope | | | | | | |
| TIA/Stroke/SE | | | | | | |
| ACS (UA/MI) | | | | | | |
| Rate/Rhythm | | | | | | |
| Stroke | | | | | | |
| Ischemic | | | | | | |
| Other | | | | | | |
| All-cause mortality | | | | | | |

Table 4a: Sensitivity analysis using commonly used patient-level methods such as random-intercept model and meta-analytic cluster-level methods.

| Outcome<br>(Usual Care is reference) | Random-<br>intercept model<br>HR (95% CI), p-<br>value |
|---|---|
| Primary | |
| AF related ED visits or | |
| CV hospitalizations | |
| Secondary | |
| AF related ED visits | |
| Unplanned CV hospitalization | |

### Table 5a Subgroup analysis and subgroup sensitivity analyses of primary efficacy composite Outcome

| Sub-Group | HR (95% CI), Interaction term | IRR (95% CI), |
|---|---|---|
| (Usual Care is reference) | p-value | Interaction term p-<br>value |
| Practice Location | | |
| Rural | | |
| Urban | | |
| Patient Sex | | |
| Female | | |
| Male | | |
| Age (years) | | |
| <75 | | |
| ≥ 75 | | |
| CHADS2 | | |
| 0 | | |
| ≥1 | | |
| CHADS-VASC | | |
| 0 | | |
| ≥ 1 | | |
| Hypertension | | |
| Yes | | |
| No | | |
| Diabetes | | |
| Yes | | |
| No | | |
| Antithrombotics (baseline) | | |
| Yes | | |
| No | | |

## Table 5b Subgroup analysis and subgroup sensitivity analyses of the number of AF Related ED Visits

| Sub-Group | HR (95% CI), Interaction | IRR (95% CI), |
|---|---|---|
| (Usual Care is reference) | term p-value | Interaction term p-value |
| Practice Location | | |
| Rural | | |
| Urban | | |
| Patient Sex | | |
| Female | | |
| Male | | |
| Age (years) | | |
| <75 | | |
| ≥ 75 | | |
| CHADS2 | | |
| 0 | | |
| ≥1 | | |
| CHADS-VASC | | |
| 0 | | |
| ≥1 | | |
| Hypertension | | |
| Yes | | |
| No | | |
| Diabetes | | |
| Yes | | |
| No | | |
| Antithrombotics (baseline) | | |
| Yes | | |
| No | | |

Table 5c Subgroup analysis and subgroup sensitivity analyses of number of CV Hospitalizations

| Sub-Group | HR (95% CI), Interaction | IRR (95% CI), |
|---|---|---|
| (Usual Care is reference) | term p-value | Interaction term p-value |
| Practice Location | | |
| Rural | | |
| Urban | | |
| Patient Sex | | |
| Female | | |
| Male | | |
| Age (years) | | |
| <75 | | |
| ≥ 75 | | |
| CHADS2 | | |
| 0 | | |
| ≥1 | | |
| CHADS-VASC* | | |
| 0 | | |
| ≥1 | | |
| Hypertension | | |
| Yes | | |
| No | | |
| Diabetes | | |
| Yes | | |
| No | | |
| Antithrombotics (baseline) | | |
| Yes | | |
| No | | |